CLINICAL TRIAL: NCT04302493
Title: Mindfulness Matters: The Impact of Mindfulness Based Stress Reduction on Post-Stroke Cognition
Brief Title: Mindfulness Based Stress Reduction and Post-Stroke Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland, College Park (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00242665
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Stroke Sequelae; Depression; Cognitive Impairment
MeSH Terms: conditions — Stroke; Depression; Cognitive Dysfunction | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to an 8 week Mindfulness Based Stress Reduction (MBSR) course versus a traditional Stroke Support Group (SSG)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) (Experimental): Participants randomized to the MBSR arm will undergo a standard 8 week course.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Stroke Support Group (SSG) (Active Comparator): As a control group, participants will participate in 8 weeks of weekly Stroke Support Group.
  Interventions: Behavioral: Stroke Support Group (SSG)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — Participants randomized to the MBSR arm will undergo a standard 8 week course of MBSR taught by a psychologist trained in the MBSR protocol and encouraged to engage in additional individual mindfulness sessions using a cell phone application.
  Arms: Mindfulness Based Stress Reduction (MBSR)
Behavioral: Stroke Support Group (SSG) — As a control group, participants randomized to the SSG arm will participate in 8 weeks of weekly Stroke Support Group sessions to experience activity and socialization without additional mindfulness training.
  Arms: Stroke Support Group (SSG)

SUMMARY:
The investigators don't fully understand how, regardless of the size or location in the brain, minor strokes can result in significant problems with focus, attention, and multi-tasking that prevent individuals from returning to an active lifestyle, and negatively impact quality of life; but the investigators' preliminary data using magnetoencephalography (MEG) suggest that there may be disruption of the neuronal network and abnormal frontal lobe activity in the brain after stroke. Mindfulness Based Stress Reduction (MBSR) is effective at treating frontal lobe dysfunction in the form of anxiety and depression occurring during the chronic phase of stroke recovery. The aim of this study is to use MBSR to improve other forms of frontal lobe dysfunction (cognitive outcomes) during the subacute phase of recovery, when patients are making critical decisions regarding patients' ability to return to work or live independently; and to use MEG, a tool capable of imaging brain activity and neuronal networks, to understand the brain changes that correspond to improvement after treatment.

DETAILED DESCRIPTION:
Thrombectomy has significantly improved stroke outcomes. Nearly 80% of the investigators' clinic population now present with small strokes and low NIH Stroke Scale (NIHSS) scores. However, despite "good recoveries", greater than 40% endorse significant problems with concentration, attention, executive function, processing speed, and mood during the subacute phase of recovery. This dysfunction prohibits individuals from fully reintegrating into the individuals' prior home and workplace environments and can result in early retirement or loss of independence, particularly in the older population. Some degree of recovery is observed by 6 months, but it is often incomplete or too late to reverse prior life-altering decisions. The impaired executive function and processing speed appear to occur independent of stroke size, location, or co-existing depression.

Magnetoencephalography (MEG) is a functional imaging tool able to evaluate neurophysiologic processes in real time similar to EEG, but with better spatial resolution. The investigators' prior work with MEG suggests that cerebral activation patterns are not only slowed and more dispersed during task completion in individuals with minor stroke compared to controls, but that there is abnormal activity in the frontal lobes, even at rest. Unfortunately, many patients do not qualify for rehabilitation and there is little data regarding effective treatment options to hasten or augment recovery.

Mindfulness training may provide an attractive therapeutic option. A combination of meditation, body awareness, and yoga, Mindfulness Based Stress Reduction (MBSR) is an active process thought to engage the frontal lobes. MBSR has been shown to improve anxiety and depression in patients with chronic disease states like migraine and diabetes, and has also been evaluated in a small series of patients with chronic stroke and traumatic brain injury demonstrating improved performance during tasks of executive function.

The investigators propose to study the effect of MBSR in the early phase of stroke recovery to determine if this intervention can help to prevent post-stroke morbidity. A cohort of patients [NIHSS <8, modified Rankin Scale (mRS) 0-2] will be enrolled. Half will be randomized to a standard 8 week course of MBSR, while the control group will instead participate in a weekly Stroke Support Group (SSG). Depression, cognition, patient perception of recovery, and degree of re-integration into prior environments will be evaluated pre- and post-intervention to determine the impact of mindfulness training on subacute post-stroke depression and cognition. All participants will undergo neuroimaging using MEG pre- and post-intervention to determine the neurophysiologic effect of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) presenting with neurological symptoms due to acute ischemic stroke (symptom onset within the week prior to admission).
* Evidence on brain MRI of acute ischemic stroke (imaging negative strokes and transient ischemic attacks (TIAs) will be excluded).
* Native English speaker (by self-report) prior to stroke.
* NIHSS <8 at initial follow-up visit (approximately 30 days post-stroke).
* mRS 0-2 at initial follow-up visit.

Exclusion Criteria:

* Primary intracerebral hemorrhage- as evidenced by blood on head CT or MRI.
* Presence of proximal large vessel occlusion.
* Cortical exam findings including aphasia or neglect.
* Prior history of dementia or undertreated psychiatric illness.
* Uncorrected hearing or visual loss.
* Inability to attend weekly MBSR or Stroke Support Group sessions.
* Inability to travel to College Park (UMD) for 2 MEG recording sessions.
* Presence of any of the following that would lead to significant artifact on MEG: cardiac pacemaker, intracranial clips, metal implants or external clips within 10mm of the head, metal implants in the eyes (unlikely given that all patients will have an MRI and criteria are similar).
* Claustrophobia, obesity, and/or any other reason leading to difficulty staying in the MEG machine for up to 1 hour.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Marsh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon request of the PI. Otherwise, de-identified results will be reported in aggregate.
Supporting Information: Study Protocol, SAP
Time Frame: Results will be published at the conclusion of the study.
Access Criteria: Upon request

REFERENCES:
- [Background] Chen K, Marsh EB. Chronic post-stroke fatigue: It may no longer be about the stroke itself. Clin Neurol Neurosurg. 2018 Nov;174:192-197. doi: 10.1016/j.clineuro.2018.09.027. Epub 2018 Sep 17. PMID 30266010
- [Background] Marsh EB, Lawrence E, Hillis AE, Chen K, Gottesman RF, Llinas RH. Pre-stroke employment results in better patient-reported outcomes after minor stroke: Short title: Functional outcomes after minor stroke. Clin Neurol Neurosurg. 2018 Feb;165:38-42. doi: 10.1016/j.clineuro.2017.12.020. Epub 2017 Dec 27. PMID 29306185
- [Background] Marsh EB, Lawrence E, Gottesman RF, Llinas RH. The NIH Stroke Scale Has Limited Utility in Accurate Daily Monitoring of Neurologic Status. Neurohospitalist. 2016 Jul;6(3):97-101. doi: 10.1177/1941874415619964. Epub 2015 Dec 13. PMID 27366291
- [Result] Girgenti SG, Dallasta I, Lawrence E, Merbach D, Simon JZ, Llinas RH, Gould NF, Marsh EB. Modified-mindfulness-based stress reduction as a treatment for cognitive recovery in patients with minor stroke: a randomized controlled pilot study. Front Neurol. 2025 Aug 26;16:1534480. doi: 10.3389/fneur.2025.1534480. eCollection 2025. PMID 40933043
- See also: Marsh Lab Website — http://marshlab.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
Started | 16 | 14
Completed | 14 | 14
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG) | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.7) | 63.6 (17.2) | 64.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30
Education [Mean (Standard Deviation); unit: years] | 12.8 (1.8) | 14.6 (3.2) | 13.5 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition as Assessed by the Montreal Cognitive Assessment Score
Description: The Montreal Cognitive Assessment (MoCA) tests executive function, attention, concentration, memory, and processing speed. The MoCA is scored on a scale of 0-30. Scores of less than 26 are considered abnormal.
Time Frame: Pre-intervention (1 month post-stroke) and post-intervention visit (6 months post-stroke)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
Number analyzed (Participants) | 14 | 14
score on a scale
  1 month | 23.5 (5.2) | 22.5 (5.9)
  6 months | 25.5 (3.7) | 23.7 (6.0)

2. Primary Outcome: Change in Cerebral Activity as Assessed by Functional Connectivity on Magnetoencephalography (MEG)
Description: Participants will undergo an MEG evaluating functional connectivity during resting state.
  GC links within the ipsilesional FPC were determined and differences in link count is reported below.
Time Frame: Pre-intervention (1 month post-stroke) and post-intervention visit (6 months post-stroke)
Population: 21 patients returned and successfully completed their follow-up MEG leaving 21 pairs of MEG data for analysis of this outcome.
Measure: Mean (Standard Error); unit: GC links
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
Number analyzed (Participants) | 13 | 8
GC links
  1 month | 1.99 (0.83) | 0 (0)
  6 months | 2.19 (0.90) | 0 (0)

3. Primary Outcome: Change in Quality of Life as Assessed by a Likert Scale
Description: Patient-reported assessment of quality of life (Likert scale 1-7 with 7 being a better QOL) at the 1 and 6 month visits. Mean of participant choice is reported.
Time Frame: Pre-intervention (1 month post-stroke) and post-intervention visit (6 months post-stroke)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
Number analyzed (Participants) | 14 | 14
score on a scale
  1 month | 5.7 (2.2) | 6.1 (1.1)
  6 months | 5.2 (1.9) | 5.1 (1.8)

4. Primary Outcome: Change in Depression as Assessed by the Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 will be administered to participants to evaluate for post-stroke depression. The PHQ-9 is scored on a scale of 0-27 with scores of 5-9 being indicative of mild depression and higher scores more severe depression.
Time Frame: Pre-intervention (1 months post-stroke) and post-intervention visit (6 months post-stroke)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
Number analyzed (Participants) | 14 | 14
score on a scale
  1 month | 6.7 (7.3) | 5.2 (5.9)
  6 months | 6.1 (6.9) | 4.9 (3.9)

ADVERSE EVENTS:
Time Frame: Up to 6 months.
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Stroke Support Group (SSG)
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
9 participants either did not complete the second MEG visit or had technical difficulties, resulting in only 21 pairs of pre- and post-MEG data available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04302493/Prot_SAP_000.pdf